CLINICAL TRIAL: NCT00945139
Title: Phase II Study of Bevacizumab and Doxil in the Treatment of Platinum-Resistant or Refractory Ovarian Cancer
Brief Title: Study of Bevacizumab/Doxil in Treatment of Platinum-Resistant/Refractory Ovarian Cancer (CA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Genentech, Inc. (Industry); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST AVF3911s; NCI-2011-02890 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; Doxorubicin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm: Doxil and Avastin (Experimental): Patients receive both agents, doxil and Avastin.
  Interventions: Drug: Doxil; Drug: Avastin

INTERVENTIONS:
Drug: Doxil — Open label study of Doxil given as 30 mg/m2 every three weeks by itself in cycle 1
  Other Names: Doxorubicin
Drug: Avastin — First agent (Doxil) will be following by Avastin 15 mg/kg on cycle 2 and every cycle thereafter until disease progression
  Other Names: Bevacizumab

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of two chemotherapy drugs, pegylated liposomal doxorubicin (Doxil) and bevacizumab (Avastin). How Doxil is metabolized and excreted from the body will also be studied.

DETAILED DESCRIPTION:
Avastin:

Avastin is a humanized monoclonal antibody (a type of protein that is normally made by the immune system to help defend the body from infection and cancer). Avastin has been approved for the treatment of colorectal cancer and lung cancer. Avastin is investigational for the treatment of ovarian cancer and has not been approved by the United States Food and Drug Administration (FDA) for this use.

Avastin is thought to work by attaching to a protein called vascular endothelial growth factor (VEGF) to block its action. VEGF plays a role in the formation of both normal and abnormal blood vessels. It is present in normal tissues, but is produced in excess by most solid cancers (tumors). In cancer, VEGF helps blood vessels bring nutrients to tumor cells, allowing the tumor cells to grow. In laboratory studies with human cancer cells grown in animals, Avastin has been shown to prevent or slow the growth of different types of cancer cells by blocking the effects of VEGF.

Doxorubicin:

Doxorubicin is a type of antibiotic that is only used in cancer chemotherapy. It slows or stops the growth of cancer. Doxorubicin has been approved by the FDA to treat cancers of the head, neck, cervix, vagina, testes, prostate, uterus and Ewing's tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be platinum resistant
* Patients will be included in the study based on the following criteria:

  * No prior anthracycline use
  * PS less or equal 2
  * Lab values within certain limits (ANC greater 1000, platelets greater 100,000; ALT, AST 2 time ULN, creatinine less 2.0)
  * No more than 3 prior chemotherapy regimens, only 2 of which can have included platinum-containing regimens
  * Use of effective means of contraception in subjects of child-bearing potential

Exclusion Criteria:

1. Disease-Specific Exclusions:

   * Evidence of complete or partial bowel obstruction
   * Need for IV hydration or TPN
   * Greater 2 prior abdominal surgeries
   * History of gastrointestinal perforation
   * Gastrointestinal perforation due to any other cause within the last 6 months
2. General Medical Exclusions:

   * Inability to comply with study and/or follow-up procedures
   * Life expectancy of less than 12 weeks
   * Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
3. Avastin-Specific Exclusions

   * Inadequately controlled hypertension (defined as systolic blood pressure 150 and/or diastolic blood pressure greater 100 mmHg on antihypertensive medications)
   * Any prior history of hypertensive crisis or hypertensive encephalopathy
   * New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
   * History of myocardial infarction or unstable angina within 6 months prior to study enrollment
   * History of stroke or transient ischemic attack within 6 months prior to study enrollment
   * Known CNS disease
   * Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
   * Symptomatic peripheral vascular disease
   * Evidence of bleeding diathesis or coagulopathy
   * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
   * Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
   * History of abdominal fistula, or intra-abdominal abscess within 6 months prior to study enrollment
   * Serious, non-healing wound, ulcer, or bone fracture
   * Proteinuria at screening as demonstrated by either:

     * Urine protein:creatinine (UPC) ratio 1.0 at screening OR
     * Urine dipstick for proteinuria greater or equal 2plus (patients discovered to have greater or equal 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate less or equal 1g of protein in 24 hours to be eligible)
   * Known hypersensitivity to any component of Avastin
   * Pregnant (positive pregnancy test) or lactating. No effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire F. Verschraegen, M.D., Principal Investigator — University of New Mexico; Franco Muggia, MD, Study Director — New York University Cancer Institute
Locations (3):
- United States (3):
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York University Cancer Institute, New York, New York

REFERENCES:
- [Result] Verschraegen CF, Czok S, Muller CY, Boyd L, Lee SJ, Rutledge T, Blank S, Pothuri B, Eberhardt S, Muggia F. Phase II study of bevacizumab with liposomal doxorubicin for patients with platinum- and taxane-resistant ovarian cancer. Ann Oncol. 2012 Dec;23(12):3104-3110. doi: 10.1093/annonc/mds172. Epub 2012 Jul 31. PMID 22851407
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 patients were screened for this study at all sites beginning March 2007. 46 patients were enrolled at the UNM Cancer Center, NYU Medical Center and NM Cancer Care Associates/Santa Fe.
Groups:
- Doxil (PLD) + Avastin (Bevacizumab): Open label study of Doxil given as 30 mg/m2 every three weeks by itself in cycle 1, and then followed by Avastin 15 mg/kg on cycle 2 and every cycle thereafter until disease progression (Progression-Free Survival determination) or withdrawal for other causes (unacceptable toxicity, patient preference). Patients undergoing PK determinations will have the dose of Avastin on cycle 2 given 24 hours after Doxil.
Period: Overall Study
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by RECIST Criteria
Description: Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by hysical exam and/or computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 25 months
Population: 43 out of 46 enrolled patients were assessable for PFS by RECIST criteria. The remaining patients could not be evaluated for this endpoint because of missed imaging scans that prevented analysis according to the defined criteria.
Measure: Median (Full Range); unit: Months
Groups:
- Doxil (PLD) + Avastin (Bevacizumab): Treatment was administered every 3 weeks (bevacizumab 15 mg/kg beginning on cycle 2 and PLD 30 mg/m2).
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 43
Months | 7.8 [2 to 13.3]

2. Secondary Outcome: Overall Survival
Description: The time from treatment initiation to death by any cause
Time Frame: 4 years
Measure: Median (Full Range); unit: Months
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 46
Months | 33.2 [3 to 37.5]

3. Secondary Outcome: Overall Response Rate (ORR) by RECIST
Description: ORR is the sum of the percentages of patients achieving complete and partial responses. Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 43
Percentage of participants
  Complete Response (CR) | 9 [3 to 22]
  Partial Response (PR) | 21 [10 to 36]
  Overall Response Rate (ORR) | 30 [17 to 46]

4. Secondary Outcome: Clinical Benefit Rate (by RECIST)
Description: Clinical Benefit Rate (CBR) is the sum of the percentages of patients achieving complete response, partial response, and stable disease. Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by physical exam and/or computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 43
percentage of participants
  Complete Response (CR) | 9 [3 to 22]
  Partial Response (PR) | 21 [10 to 36]
  Stable Disease (SD) | 56 [40 to 71]
  Clinical Benefit Rate (CBR) | 86 [72 to 95]

5. Secondary Outcome: Overall Response Rate (ORR) by GCIC Criteria
Description: A response according to GCIC criteria has occurred if there is at least a 50% reduction in CA 125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA-125 only if they have a pretreatment sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 28
percentage of participants | 50 [31 to 69]

6. Primary Outcome: Progression Free Survival (PFS) by GCIC Criteria
Description: Using GCIC criteria, progression is defined as CA-125 levels greater than, or equal to, 2 times the upper limit of a reference range on 2 occasions and at least 1 week apart.
Time Frame: Up to 25 months
Population: 28 out of 46 enrolled patients were assessable for PFS per GCIC criteria. The remaining patients could not be evaluated for this endpoint because the timing of their CA-125 measurements did not meet the defined criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Number analyzed (Participants) | 28
Months | 6.6 [1 to 24.6]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Doxil (PLD) + Avastin (Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxil (PLD) + Avastin (Bevacizumab) (N=46)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Speech impairment: global aphasia (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagoscopy abnormal: ulceration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxil (PLD) + Avastin (Bevacizumab) (N=46)
Allergic reaction (General disorders) | 4 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (9)
Leukocyte count decreased (Blood and lymphatic system disorders) | 5 (11)
Neutrophil count decreased (Blood and lymphatic system disorders) | 6 (8)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (7)
Hypertension (High blood pressure) (Cardiac disorders) | 18 (34)
Fatigue (General disorders) | 23 (40)
Fever (General disorders) | 3 (3)
Weight Loss (Metabolism and nutrition disorders) | 5 (7)
Skin disorders - Other (Skin and subcutaneous tissue disorders) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (13)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 21 (76)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 15 (22)
Desquamating rash (Skin and subcutaneous tissue disorders) | 5 (9)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 14 (20)
Constipation (Gastrointestinal disorders) | 15 (22)
Diarrhea (Gastrointestinal disorders) | 8 (13)
Dyspepsia (Indigestion) (Gastrointestinal disorders) | 3 (4)
Mucositis - oral (Mouth inflammation) (Gastrointestinal disorders) | 9 (16)
Nausea (Gastrointestinal disorders) | 17 (32)
Vomiting (Gastrointestinal disorders) | 6 (12)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 8 (11)
Dehydration (Gastrointestinal disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (8)
Edema: limbs (General disorders) | 4 (5)
Hyperglycemia (High blood glucose) (Investigations) | 9 (17)
Hypocalcemia (Low calcium levels) (Investigations) | 4 (4)
Hypokalemia (Low potassium levels) (Investigations) | 5 (8)
Hypomagnesemia (Low magnesium levels) (Investigations) | 3 (5)
Hyponatremia (Low sodium levels) (Investigations) | 8 (13)
Creatinine increased (Investigations) | 5 (8)
Proteinuria (Investigations) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Muscle pain) (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Pain - Other (Musculoskeletal and connective tissue disorders) | 8 (9)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 20 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (15)
Anxiety (Nervous system disorders) | 5 (6)
Depression (Nervous system disorders) | 3 (3)
Blurred vision (Eye disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Nosebleed) (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Ear, nose and throat examination abnormal (General disorders) | 14 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No